CLINICAL TRIAL: NCT04342819
Title: The Effect of empagliFlozin on Platelet Function profilEs in diabetiC patienTs - The EFFECT Study.
Acronym: EFFECT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The University of The West Indies (Other)
Responsible Party: Principal Investigator, Naveen Seecheran, Principal Investigator, The University of The West Indies
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CREC-SA.0054/10/2019
Record Dates: First submitted 2020-04-08; First posted 2020-04-13 (Actual); Results first posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Platelet Dysfunction Due to Drugs
MeSH Terms: interventions — Sodium-Glucose Transporter 2 Inhibitors; empagliflozin

STUDY DESIGN:
Intervention Model Description: The study will be of a prospective, single-arm, crossover trial design over a 2-year period. Patients at the Eric Williams Medical Sciences Complex (EWMSC), Mt. Hope, Trinidad and Tobago.
Masking Description: Open-Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- SGLT2i (Experimental): Empagliflozin 25 mg per oral once daily
  Interventions: Drug: SGLT2 inhibitor

INTERVENTIONS:
Drug: SGLT2 inhibitor — Sodium-Glucose Like Transporter 2 Inhibitor
  Other Names: Empagliflozin

SUMMARY:
The mechanistic effects of empagliflozin on platelet function profiles have not yet been ascertained.

DETAILED DESCRIPTION:
Sodium GLucose Transport 2 inhibitors (SGLT2I), including empagliflozin, reduce the likelihood of hospitalization for heart failure and death in persons with type 2 diabetes, of which the mechanism has not been fully elucidated. The mechanistic effects of empagliflozin on platelet function profiles have not yet been ascertained. It remains unclear if this reduction in cardiovascular death is mediated by decreased platelet reactivity.

ELIGIBILITY:
Inclusion Criteria:

1. between 18 and 74 years of age,
2. have stable coronary artery disease and diabetes mellitus, already on DAPT with aspirin and clopidogrel for at least 6 months,

Exclusion Criteria:

1. presence of active internal bleeding or history of bleeding diathesis or clinical findings associated with an increased risk of bleeding,
2. history of ischemic or hemorrhagic stroke, transient ischemic attack, intracranial neoplasm, arteriovenous malformation, or aneurysm,
3. history of clinical and/or hemodynamic instability,
4. within 1 month of placement of a bare metal stent,
5. within 30 days of coronary artery bypass graft surgery or PCI without a stent placed,
6. planned coronary revascularization,
7. treatment with fibrin-specific fibrinolytic therapy <24 h or non-fibrin-specific fibrinolytic therapy <48 h,
8. use of an oral anticoagulation agent or international normalized ratio >1.5,
9. body weight <60 kg,
10. age >75 years,
11. hemoglobin <10 g/dL,
12. platelet count <100×106/μL,
13. creatinine >2 mg/dL,
14. hepatic enzymes >2.5 times the upper limit of normal,
15. pregnancy and/or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Eric Williams Medical Sciences Complex, Port of Spain, North, Trinidad and Tobago

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Seecheran N, Ramdeen A, Debideen N, Ali K, Grimaldos K, Grimaldos G, Karan A, Seecheran R, Seecheran V, Persad S, Abdullah H, Peram L, Giddings S, Motilal S, Tello-Montoliu A, Schneider D. The Effect of Empagliflozin on Platelet Function Profiles in Patients with Stable Coronary Artery Disease in Trinidad: The EFFECT Pilot Study. Cardiol Ther. 2021 Jun;10(1):189-199. doi: 10.1007/s40119-020-00208-0. Epub 2020 Dec 11. PMID 33306161

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants provided written informed consent to participate in this prospective, open-label study that aimed to assess the effect of empagliflozin 25 mg once daily for 10 days. Patients were screened and enrolled between January 2020 and August 2020 at the cardiology outpatient clinic at our institution (Eric Williams Medical Sciences Complex, Trinidad and Tobago).
Pre-assignment Details: No enrolled patients were excluded from the study before assignment to empagliflozin.
Period: Overall Study
Arm/Group | SGLT2i
Started | 25
Completed | 20
Not Completed | 5
Not completed — Declined | 4
Not completed — Not meeeting selection criteria | 1

BASELINE CHARACTERISTICS:
Arm/Group | SGLT2i
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.2 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 19
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Trinidad and Tobago | 100
P2Y12 Reaction Units (PRU) [Mean (Standard Deviation); unit: P2Y12 Reaction Units (PRU)] | 187.35 (1)

OUTCOME MEASURES:

1. Primary Outcome: P2Y12 Reaction Units
Description: P2Y12 Reaction Units post-Empagliflozin. Citrated blood samples are processed by CRAs and study investigators. The platelet function assay to be utilized is the VerifyNow P2Y12 (VN-P2Y12) assay (Accriva, San Diego, California). In brief, the VN-P2Y12 assay is a rapid whole blood point-of-care device that reports results as P2Y12 reaction units (PRU) and percent inhibition of platelet aggregation (%IPA). Assays will be performed as per the instructions of the manufacturer previously described.
Time Frame: 14 days
Measure: Mean (95% Confidence Interval); unit: P2Y12 Reaction Units
Arm/Group | SGLT2i
Number analyzed (Participants) | 20
P2Y12 Reaction Units | 187.35 [155.38 to 219.32]

ADVERSE EVENTS:
Time Frame: 28 days.
Arm/Group | SGLT2i
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-01): https://cdn.clinicaltrials.gov/large-docs/19/NCT04342819/Prot_SAP_001.pdf